CLINICAL TRIAL: NCT03900117
Title: Hypofractionated Radiotherapy Followed by Hypofractionated Boost With Weekly Concurrent Chemotherapy for Unresectable Stage III Non-Small Cell Lung Cancer: A Prospective, Single Arm Phase II Study
Brief Title: Hypofractionated Radiotherapy Followed by Hypo-boost for Local Advanced NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO 1049
Record Dates: First submitted 2019-03-31; First posted 2019-04-02 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; hypofractionated radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- split-course radiotherapy (Experimental): The radiotherapy is delivered using simultaneous integrated boost (SIB)-intensity-modulated radiotherapy (IMRT). Patients are irradiation at a palliative dose at the initial course: 40Gy/10f to gross tumor. The disease is re-evaluated one month after the end of the initial course using CT. The patient who achieved a partial remission according to the RECIST criteria and had a recovery of lung function should get the additional boost. At the second course, the tumor is re-simulated. The residual tumor was then treated with the second course of radiotherapy. A dose of 28Gy/7f is delivered to the residue tumor. Concurrent chemotherapy consists of weekly docetaxel(25mg/㎡) and nedaplatin(25mg/㎡), each of 1 day's duration.
  Interventions: Radiation: split-course radiotherapy; Drug: concurrent chemotherapy

INTERVENTIONS:
Radiation: split-course radiotherapy — Patients are irradiation at a palliative dose at the initial course: 40Gy/10f to PTV-GTV. The disease is re-evaluated one month after the end of the initial course using CT. The patient who achieved a partial remission according to the RECIST criteria and had a recovery of lung function should get the additional boost. At the second course, the tumor is repositioned and scanned. The residual tumor was then treated with the second course of radiotherapy. A dose of 28Gy/7f is delivered to the residue tumor.
Drug: concurrent chemotherapy — Concurrent chemotherapy consists of weekly docetaxel(25mg/㎡) and nedaplatin(25mg/㎡), each of 1 day's duration.

SUMMARY:
The primary objective is to assess the safety and efficacy of hypofractionated radiotherapy followed by hypo-boost combined with concurrent weekly chemotherapy in unresectable LA-NSCLC patients.

DETAILED DESCRIPTION:
Patients receive four cycles of weekly docetaxel(25mg/㎡) and nedaplatin(25mg/㎡), each of 1 day's duration, concurrent with split-course thoracic radiotherapy of 40 Gy/10 fractions and 28 Gy/7 fractions administered in the first and second courses, respectively, with one-month break. The primary end point is progression-free survival, which is the time that passes from the first day of radiotherapy to the date at which disease progresses. Progression-free survival will be calculated using the Kaplan-Meier method.Toxicities will be graded according to CTCAE v. 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of NSCLC.
* Patients have measurable or evaluable lesions based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Unresectable phase IIIA(N2) and IIIB lung cancer confirmed by PET/CT, CT or MRI.
* Whole lung V20>=35% when giving 60Gy which is the minimum dose of radical irradiation.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Previously treated with chemotherapy or treatment-naive
* No previous chest radiotherapy, immunotherapy or biotherapy
* Hemoglobin≥10 mg/dL, platelet≥100000/μL,absolute neutrophil count ≥1500/μL
* Serum creatinine ≤1.25 times the upper normal limit(UNL), or creatinine clearance≥60 ml/min
* Bilirubin ≤1.5 times UNL, AST（SGOT）≤2.5 times UNL ,ALT（SGPT）≤2.5 times UNL,alkaline phosphatase ≤5 times UNL
* FEV1 >0.8 L
* CB6 within normal limits
* patients and their family signed the informed consents

Exclusion Criteria:

* Previous or recent another malignancy, except nonmelanoma skin cancer or cervical cancer in situ
* Contraindication for chemotherapy
* Malignant pleural or pericardial effusion.
* Women in pregnancy, lactation period, or no pregnancy test 14 days before the first dose
* Women who has the probability of pregnancy without contraception
* Tendency of hemorrhage
* In other clinical trials within 30 days
* Addicted in drugs or alcohol, AIDS patients
* Uncontrollable seizure or psychotic patients without self-control ability
* Severe allergy or idiosyncrasy
* Not suitable for this study judged by researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 3 years

SECONDARY OUTCOMES:
overall survival | 3 years
response rate | 2 months
rate of grade 3-4 radiation esophagitis | 1 year
rate of grade 3-4 radiation pneumonitis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Hui Liu, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Schrum D, Carter D, Kelsey C, et al: Non Small Cell Lung Cancer (ed 9). Philadelphia, PA, Lippincott Williams & Wilkins, 2011, pp 799-847.
- [Background] Dillman RO, Seagren SL, Propert KJ, Guerra J, Eaton WL, Perry MC, Carey RW, Frei EF 3rd, Green MR. A randomized trial of induction chemotherapy plus high-dose radiation versus radiation alone in stage III non-small-cell lung cancer. N Engl J Med. 1990 Oct 4;323(14):940-5. doi: 10.1056/NEJM199010043231403. PMID 2169587
- [Background] Sause W, Kolesar P, Taylor S IV, Johnson D, Livingston R, Komaki R, Emami B, Curran W Jr, Byhardt R, Dar AR, Turrisi A 3rd. Final results of phase III trial in regionally advanced unresectable non-small cell lung cancer: Radiation Therapy Oncology Group, Eastern Cooperative Oncology Group, and Southwest Oncology Group. Chest. 2000 Feb;117(2):358-64. doi: 10.1378/chest.117.2.358. PMID 10669675
- [Background] Curran WJ, Scott C, Langer C, et al. Phase III comparision of sequential vs concurrent chemoradiation therapy for patients with unresectable stage III non-small cell lung cancer: initial report of RTOG 9410. Proc Am Soc Clin Oncol, 2000, 19: 484a.
- [Background] Furuse K, Fukuoka M, Kawahara M, Nishikawa H, Takada Y, Kudoh S, Katagami N, Ariyoshi Y. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with mitomycin, vindesine, and cisplatin in unresectable stage III non-small-cell lung cancer. J Clin Oncol. 1999 Sep;17(9):2692-9. doi: 10.1200/JCO.1999.17.9.2692. PMID 10561343
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Pfister DG, Johnson DH, Azzoli CG, Sause W, Smith TJ, Baker S Jr, Olak J, Stover D, Strawn JR, Turrisi AT, Somerfield MR; American Society of Clinical Oncology. American Society of Clinical Oncology treatment of unresectable non-small-cell lung cancer guideline: update 2003. J Clin Oncol. 2004 Jan 15;22(2):330-53. doi: 10.1200/JCO.2004.09.053. Epub 2003 Dec 22. No abstract available. PMID 14691125
- [Background] Strom HH, Bremnes RM, Sundstrom SH, Helbekkmo N, Flotten O, Aasebo U. Concurrent palliative chemoradiation leads to survival and quality of life benefits in poor prognosis stage III non-small-cell lung cancer: a randomised trial by the Norwegian Lung Cancer Study Group. Br J Cancer. 2013 Sep 17;109(6):1467-75. doi: 10.1038/bjc.2013.466. Epub 2013 Aug 20. PMID 23963145
- [Background] Strom HH, Bremnes RM, Sundstrom SH, Helbekkmo N, Aasebo U. Poor prognosis patients with inoperable locally advanced NSCLC and large tumors benefit from palliative chemoradiotherapy: a subset analysis from a randomized clinical phase III trial. J Thorac Oncol. 2014 Jun;9(6):825-33. doi: 10.1097/JTO.0000000000000184. PMID 24807158
- [Background] Lau DH, Crowley JJ, Gandara DR, Hazuka MB, Albain KS, Leigh B, Fletcher WS, Lanier KS, Keiser WL, Livingston RB. Southwest Oncology Group phase II trial of concurrent carboplatin, etoposide, and radiation for poor-risk stage III non-small-cell lung cancer. J Clin Oncol. 1998 Sep;16(9):3078-81. doi: 10.1200/JCO.1998.16.9.3078. PMID 9738578
- [Background] Davies AM, Chansky K, Lau DH, Leigh BR, Gaspar LE, Weiss GR, Wozniak AJ, Crowley JJ, Gandara DR; SWOG S9712. Phase II study of consolidation paclitaxel after concurrent chemoradiation in poor-risk stage III non-small-cell lung cancer: SWOG S9712. J Clin Oncol. 2006 Nov 20;24(33):5242-6. doi: 10.1200/JCO.2006.07.0268. PMID 17114656
- [Background] Robnett TJ, Machtay M, Vines EF, McKenna MG, Algazy KM, McKenna WG. Factors predicting severe radiation pneumonitis in patients receiving definitive chemoradiation for lung cancer. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):89-94. doi: 10.1016/s0360-3016(00)00648-9. PMID 10924976
- [Background] Torre-Bouscoulet L, Munoz-Montano WR, Martinez-Briseno D, Lozano-Ruiz FJ, Fernandez-Plata R, Beck-Magana JA, Garcia-Sancho C, Guzman-Barragan A, Vergara E, Blake-Cerda M, Gochicoa-Rangel L, Maldonado F, Arroyo-Hernandez M, Arrieta O. Abnormal pulmonary function tests predict the development of radiation-induced pneumonitis in advanced non-small cell lung Cancer. Respir Res. 2018 Apr 24;19(1):72. doi: 10.1186/s12931-018-0775-2. PMID 29690880
- [Background] Wang D, Zhu J, Sun J, Li B, Wang Z, Wei L, Yin Y, Sun H, Fu Z, Zhang X, Huo Z. Functional and biologic metrics for predicting radiation pneumonitis in locally advanced non-small cell lung cancer patients treated with chemoradiotherapy. Clin Transl Oncol. 2012 Dec;14(12):943-52. doi: 10.1007/s12094-012-0890-3. Epub 2012 Jul 20. PMID 22855174
- [Background] Dehing-Oberije C, De Ruysscher D, van Baardwijk A, Yu S, Rao B, Lambin P. The importance of patient characteristics for the prediction of radiation-induced lung toxicity. Radiother Oncol. 2009 Jun;91(3):421-6. doi: 10.1016/j.radonc.2008.12.002. Epub 2009 Jan 13. PMID 19147245
- [Background] Chen S, Zhou S, Zhang J, Yin FF, Marks LB, Das SK. A neural network model to predict lung radiation-induced pneumonitis. Med Phys. 2007 Sep;34(9):3420-7. doi: 10.1118/1.2759601. PMID 17926943
- [Background] Kong FM, Wang S. Nondosimetric risk factors for radiation-induced lung toxicity. Semin Radiat Oncol. 2015 Apr;25(2):100-9. doi: 10.1016/j.semradonc.2014.12.003. Epub 2014 Dec 15. PMID 25771414
- [Background] Inoue A, Kunitoh H, Sekine I, Sumi M, Tokuuye K, Saijo N. Radiation pneumonitis in lung cancer patients: a retrospective study of risk factors and the long-term prognosis. Int J Radiat Oncol Biol Phys. 2001 Mar 1;49(3):649-55. doi: 10.1016/s0360-3016(00)00783-5. PMID 11172945
- [Background] Ferrero C, Badellino S, Filippi AR, Focaraccio L, Giaj Levra M, Levis M, Moretto F, Torchio R, Ricardi U, Novello S. Pulmonary function and quality of life after VMAT-based stereotactic ablative radiotherapy for early stage inoperable NSCLC: a prospective study. Lung Cancer. 2015 Sep;89(3):350-6. doi: 10.1016/j.lungcan.2015.06.019. Epub 2015 Jun 26. PMID 26164208
- [Background] Blackstock AW, Socinski MA, Bogart J, et al; Cancer and Leukemia Group B. Induction plus concurrent chemotherapy with high-dose (74 Gy) 3-dimensional (3-D) thoracic radiotherapy in stage III non-small cell lung cancer. Preliminary report of Cancer and Leukemia Group B (CALGB) 30105. Proc Am Soc Clin Oncol 2006;24(18S):Abstr 7042.
- [Background] Lee CB, Socinski A, Lin L, et al. High-dose 3D chemoradiotherapy in stage III non-small cell lung cancer (NSCLC) at the University of North Carolina: long-term follow up and late complications. Proc Am Soc Clin Oncol 2006;24(18S):Abstr 7145.
- [Background] Kong FM, Ten Haken RK, Schipper MJ, Sullivan MA, Chen M, Lopez C, Kalemkerian GP, Hayman JA. High-dose radiation improved local tumor control and overall survival in patients with inoperable/unresectable non-small-cell lung cancer: long-term results of a radiation dose escalation study. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):324-33. doi: 10.1016/j.ijrobp.2005.02.010. PMID 16168827
- [Background] Schild SE, McGinnis WL, Graham D, Hillman S, Fitch TR, Northfelt D, Garces YI, Shahidi H, Tschetter LK, Schaefer PL, Adjei A, Jett J. Results of a Phase I trial of concurrent chemotherapy and escalating doses of radiation for unresectable non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):1106-11. doi: 10.1016/j.ijrobp.2006.02.046. Epub 2006 May 26. PMID 16730134
- [Background] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Background] Hanna N, Neubauer M, Yiannoutsos C, McGarry R, Arseneau J, Ansari R, Reynolds C, Govindan R, Melnyk A, Fisher W, Richards D, Bruetman D, Anderson T, Chowhan N, Nattam S, Mantravadi P, Johnson C, Breen T, White A, Einhorn L; Hoosier Oncology Group; US Oncology. Phase III study of cisplatin, etoposide, and concurrent chest radiation with or without consolidation docetaxel in patients with inoperable stage III non-small-cell lung cancer: the Hoosier Oncology Group and U.S. Oncology. J Clin Oncol. 2008 Dec 10;26(35):5755-60. doi: 10.1200/JCO.2008.17.7840. Epub 2008 Nov 10. PMID 19001323
- [Background] Spoelstra FO, Pantarotto JR, van Sornsen de Koste JR, Slotman BJ, Senan S. Role of adaptive radiotherapy during concomitant chemoradiotherapy for lung cancer: analysis of data from a prospective clinical trial. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1092-7. doi: 10.1016/j.ijrobp.2008.12.027. Epub 2009 Mar 26. PMID 19327915
- [Background] Gielda BT, Marsh JC, Zusag TW, Faber LP, Liptay M, Basu S, Warren WH, Fidler MJ, Batus M, Abrams RA, Bonomi P. Split-course chemoradiotherapy for locally advanced non-small cell lung cancer: a single-institution experience of 144 patients. J Thorac Oncol. 2011 Jun;6(6):1079-86. doi: 10.1097/JTO.0b013e3182199a7c. PMID 21532501
- [Background] Belani CP, Choy H, Bonomi P, Scott C, Travis P, Haluschak J, Curran WJ Jr. Combined chemoradiotherapy regimens of paclitaxel and carboplatin for locally advanced non-small-cell lung cancer: a randomized phase II locally advanced multi-modality protocol. J Clin Oncol. 2005 Sep 1;23(25):5883-91. doi: 10.1200/JCO.2005.55.405. Epub 2005 Aug 8. PMID 16087941
- [Background] Curran W, Scott C, Langer C, et al. Phase III comparison of sequential vs concurrent chemoradiotherapy for patients (pts) with unresected stage III non-small cell lung cancer (NSCLC): report of Radiation Therapy Oncology Group (RTOG) 9410. Proc Am Soc Clin Oncol 2003;22:Abstr 2499.
- [Background] Albain KS, Swann RS, Rusch VW, Turrisi AT 3rd, Shepherd FA, Smith C, Chen Y, Livingston RB, Feins RH, Gandara DR, Fry WA, Darling G, Johnson DH, Green MR, Miller RC, Ley J, Sause WT, Cox JD. Radiotherapy plus chemotherapy with or without surgical resection for stage III non-small-cell lung cancer: a phase III randomised controlled trial. Lancet. 2009 Aug 1;374(9687):379-86. doi: 10.1016/S0140-6736(09)60737-6. Epub 2009 Jul 24. PMID 19632716
- [Background] Vokes EE, Herndon JE 2nd, Kelley MJ, Cicchetti MG, Ramnath N, Neill H, Atkins JN, Watson DM, Akerley W, Green MR; Cancer and Leukemia Group B. Induction chemotherapy followed by chemoradiotherapy compared with chemoradiotherapy alone for regionally advanced unresectable stage III Non-small-cell lung cancer: Cancer and Leukemia Group B. J Clin Oncol. 2007 May 1;25(13):1698-704. doi: 10.1200/JCO.2006.07.3569. Epub 2007 Apr 2. PMID 17404369
- [Background] Segawa Y, Kiura K, Takigawa N, Kamei H, Harita S, Hiraki S, Watanabe Y, Sugimoto K, Shibayama T, Yonei T, Ueoka H, Takemoto M, Kanazawa S, Takata I, Nogami N, Hotta K, Hiraki A, Tabata M, Matsuo K, Tanimoto M. Phase III trial comparing docetaxel and cisplatin combination chemotherapy with mitomycin, vindesine, and cisplatin combination chemotherapy with concurrent thoracic radiotherapy in locally advanced non-small-cell lung cancer: OLCSG 0007. J Clin Oncol. 2010 Jul 10;28(20):3299-306. doi: 10.1200/JCO.2009.24.7577. Epub 2010 Jun 7. PMID 20530281
- [Background] Fu KK, Pajak TF, Trotti A, Jones CU, Spencer SA, Phillips TL, Garden AS, Ridge JA, Cooper JS, Ang KK. A Radiation Therapy Oncology Group (RTOG) phase III randomized study to compare hyperfractionation and two variants of accelerated fractionation to standard fractionation radiotherapy for head and neck squamous cell carcinomas: first report of RTOG 9003. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):7-16. doi: 10.1016/s0360-3016(00)00663-5. PMID 10924966
- [Background] Saunders M, Dische S, Barrett A, Harvey A, Griffiths G, Palmar M. Continuous, hyperfractionated, accelerated radiotherapy (CHART) versus conventional radiotherapy in non-small cell lung cancer: mature data from the randomised multicentre trial. CHART Steering committee. Radiother Oncol. 1999 Aug;52(2):137-48. doi: 10.1016/s0167-8140(99)00087-0. PMID 10577699
- [Background] Petereit DG, Sarkaria JN, Chappell R, Fowler JF, Hartmann TJ, Kinsella TJ, Stitt JA, Thomadsen BR, Buchler DA. The adverse effect of treatment prolongation in cervical carcinoma. Int J Radiat Oncol Biol Phys. 1995 Jul 30;32(5):1301-7. doi: 10.1016/0360-3016(94)00635-X. PMID 7635769
- [Background] Begg AC, Hofland I, Van Glabekke M, et al. Predictive value of potential doubling time for radiotherapy of head and neck tumor patients: results from the EORTC cooperative trial 22851. Semin Radiat Oncol 1992;2:22-25.
- [Derived] Zhou R, Qiu B, Xiong M, Liu Y, Peng K, Luo Y, Wang D, Liu F, Chen N, Guo J, Zhang J, Huang X, Rong Y, Liu H. Hypofractionated Radiotherapy followed by Hypofractionated Boost with weekly concurrent chemotherapy for Unresectable Stage III Non-Small Cell Lung Cancer: Results of A Prospective Phase II Study (GASTO-1049). Int J Radiat Oncol Biol Phys. 2023 Oct 1;117(2):387-399. doi: 10.1016/j.ijrobp.2023.04.021. Epub 2023 Apr 25. PMID 37100160